CLINICAL TRIAL: NCT02960698
Title: Identifying the Neural Correlates of Cognitive Impulsivity in Patients With Tourette Syndrome. "COGIT".
Brief Title: Impulsivity in Tourette Syndrome : Behavioral and Neuroimaging Study
Acronym: COGIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C16-07; 2016-A00936-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-10-27; First posted 2016-11-10 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2021-08

CONDITIONS: Tourette Syndrome
Keywords: cognitive impulsivity; IRM; Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TREATED PATIENT WITH TOURETTE SYNDROME (Active Comparator): comportemental tasks included impulsivity tests will performed at V1 Resting state IRM will be performed at V2 40 patients
  Interventions: Other: IRM and comportemental tasks
- UNTREATED PATIENT WITH TOURETTE SYNDROME (Active Comparator): comportemental tasks included impulsivity tests will performed at V1 Resting state IRM will be performed at V2 40 patients
  Interventions: Other: IRM and comportemental tasks
- Healthy volunteers (Placebo Comparator): comportemental tasks included impulsivity tests will performed at V1 Resting state IRM will be performed at V2 80 subjects
  Interventions: Other: IRM and comportemental tasks

INTERVENTIONS:
Other: IRM and comportemental tasks

SUMMARY:
Tourette syndrome (TS) is characterized by the presence of multiple vocal and motor tics. Behavioral disorders associated with TS are common, particularly impulsivity, anti-sociality and socially inappropriate behavior. Specifically, cognitive impulsivity could be the source of these troubles. Its anatomical substrates is based on connections between frontal and striatal areas.

Initially, a battery of behavioral tests measuring different types of impulsivity (motor, cognitive and decision) will be administered on three groups of subjects: TS: 80 patients (40 patients treated and 40 untreated) and 40 healthy volunteers.

Then, investigators will study the fronto-striatal connections in the TS group of 80 patients (40 patients treated and 40 untreated) compared to 40 healthy volunteers using neuroimaging techniques (3T MRI). The techniques used will be functional connectivity study of "resting state" MRI (RS-fMRI) combined with a reconstruction of white matter fibers by diffusion tensor imaging (DTI). Behavioral performance will be correlated with the correlation imaging data to highlight the functional anatomical substrates of impulsivity in patients with TS.

Finally, investigators will look specifically using functional MRI activation, the anatomical and functional substrates of the three types of impulsivity (motor, cognitive and decision-making).

Through this study, investigators hope to elucidate the anatomical and functional bases of cognitive impulsivity in patients with TS and thus lay the basis for more targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* ≥ about 18 and 65 years old
* About receiving Social Security or universal health coverage or any equivalent plan
* About who signed the informed consent

For TS patients treated :

* TS principal diagnosis, based on the DSM-5 criteria
* Stable pharmacological treatment at least 4 weeks prior to study entry;
* Possibility of controlling the majority tics of the upper part of the body lying down for at least 10 minutes (frequency tics on YGTSS <3).

For TS patients untreated:

* TS principal diagnosis, based on the DSM-5 criteria
* No psychotropic treatments (neuroleptics, antidepressants or anxiolytics) mentioned at the time of inclusion.
* Possibility of controlling the majority tics of the upper part of the body lying down for at least 10 minutes (frequency tics on YGTSS <3).

In healthy volunteers:

* Normal neurological examination (evaluation MINI).
* No regular pharmacological treatment with the exception of birth control pills for women

Exclusion Criteria:

For all patients TS:

* Age <18 years.
* Presence One of the following diagnoses Axis I DSM-5: schizophrenic disorders or current psychotic episode or in the past, bipolar disorder, current major depressive disorder autism spectrum.
* Abus Psychotropic substance dependency or a psychotropic substance, including alcohol (except nicotine).
* Support Regular / chronic drugs and other xenobiotics tropic psychotropic.
* Support Treatment with benzodiazepines in the 4 months prior to study entry. -Patient Subject to a measure of legal protection (guardianship, curatorship or safeguard justice). -No private freedom by administrative decision or justice.
* No Unable to consent and are not subject to a protection measure.
* Participation In other biomedical research or subjected to an exclusion period for another search.
* Problems General understanding.
* Weight Of more than 150 kg.
* Inability To maintain an upper portion of movement of the body lying down for at least 10 minutes (frequency tics on YGTSS> 3).

In healthy volunteers (HV):

* psychiatric disorders, cognitive impairment assessed by the MINI scale.
* About not being able to understand the tasks
* age <18 years.
* No Subject to a measure of legal protection (guardianship, curatorship or safeguard justice).
* Participation In other biomedical research or subjected to an exclusion period for another search.
* Not Unable to consent and are not subject to a protection measure.
* Not private freedom by administrative decision or court

For TS patients (treated and untreated) and HV

* relative to MRI 3Tesla : pacemaker, cardiac cell or neural stimulator ferromagnetic surgical clips body intraocular or intracranial metallic foreign cochlear implant artificial heart valve or arterial metal surgical equipment metallic material that could concentrate the radio frequency pulses pregnant women, women in labor or lactating aneurism Standing up the eyelids vascular malformation of the brain
* Topic not wishing to be informed of a clinically significant abnormality discovered during the realization of MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
behavior performance (percentage of correct responses and reaction time) | up to one month
BOLD signal of functional MRI scan | up to one month

CONTACTS AND LOCATIONS:
Locations (1):
- HARTMANN, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atkinson-Clement C, de Liege A, Klein Y, Beranger B, Valabregue R, Delorme C, Roze E, Fernandez-Egea E, Hartmann A, Robbins TW, Worbe Y. The sooner the better: clinical and neural correlates of impulsive choice in Tourette disorder. Transl Psychiatry. 2021 Nov 3;11(1):560. doi: 10.1038/s41398-021-01691-2. PMID 34732691
- [Background] Atkinson-Clement C, Sofia F, Fernandez-Egea E, de Liege A, Beranger B, Klein Y, Deniau E, Roze E, Hartmann A, Worbe Y. Structural and functional abnormalities within sensori-motor and limbic networks underpin intermittent explosive symptoms in Tourette disorder. J Psychiatr Res. 2020 Jun;125:1-6. doi: 10.1016/j.jpsychires.2020.02.033. Epub 2020 Mar 4. PMID 32169732
- [Background] Atkinson-Clement C, Porte CA, de Liege A, Wattiez N, Klein Y, Beranger B, Valabregue R, Sofia F, Hartmann A, Pouget P, Worbe Y. Neural correlates and role of medication in reactive motor impulsivity in Tourette disorder. Cortex. 2020 Apr;125:60-72. doi: 10.1016/j.cortex.2019.12.007. Epub 2019 Dec 30. PMID 31978743
- [Background] Atkinson-Clement C, Porte CA, de Liege A, Klein Y, Delorme C, Beranger B, Valabregue R, Gallea C, Robbins TW, Hartmann A, Worbe Y. Impulsive prepotent actions and tics in Tourette disorder underpinned by a common neural network. Mol Psychiatry. 2021 Jul;26(7):3548-3557. doi: 10.1038/s41380-020-00890-5. Epub 2020 Sep 29. PMID 32994553